CLINICAL TRIAL: NCT04273009
Title: Percutaneous Tibial Nerve Stimulation With the Renew Anal Plug Device for the Treatment of Faecal Incontinence
Brief Title: Optimising Treatments for Faecal Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 16/LO/1821
Record Dates: First submitted 2019-02-07; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2019-02

CONDITIONS: Faecal Incontinence; Pelvic Floor Disorders
MeSH Terms: conditions — Encopresis; Pelvic Floor Disorders

STUDY DESIGN:
Intervention Model Description: Patients who have completed the treatment can switch to the other treatment offered.
Who Masked: Participant, Investigator
Masking Description: Both participants and first investigator will be masked from the actual treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Renew Anal Insert (Active Comparator): The device is intended for self-insertion through the anal canal aided by a fingertip applicator.
  Interventions: Device: Renew VS PTNS
- Percutaneous tibial nerve stimulation (Active Comparator): A fine needle is inserted next to the tibial nerve above the ankle, a ground pad is attached to the heel and electric current just strong enough to cause minor tingling is passed between these two points.
  Interventions: Device: Renew VS PTNS

INTERVENTIONS:
Device: Renew VS PTNS — These will be prescribed and applied as described above.

SUMMARY:
The purpose of the study is to directly compare two medical treatments for faecal incontinence: Renew™ Anal Insert and Percutaneous Tibial Nerve Stimulation (PTNS) for a period of 12 weeks. Both are routinely used in our practice.

DETAILED DESCRIPTION:
The Renew™ anal insert is a new single-use anal device, CE marked and widely used in the UK and Europe. It is indicated for the management of faecal incontinence and designed to seal and prevent the involuntary passage of stool from the rectum. The device is intended for self-insertion aided by a fingertip applicator.

Percutaneous tibial nerve stimulation (PTNS) is a form of electrical stimulation that offers a simple minimally invasive outpatient treatment for faecal incontinence. A fine needle is inserted next to the tibial nerve above the ankle, a ground pad is attached to the heel and electric current just strong enough to cause minor tingling is passed between these two points. The treatment requires 12 outpatients sessions that are 30 minutes long each time and the treatment may be repeated.

Patients will be randomly allocated to either receive PTNS therapy or the Renew™ device. This will be done by the investigators randomly selecting a sealed envelope that is not see-through from a large number of identical envelopes. Each of these envelopes will contain either the word PTNS or the word Renew, which will then determine patients' treatment. There will be an equal number of PTNS and Renew envelopes to make this decision truly random. The principal investigator of this study will not know which treatment patients have been allocated to until after the study is complete. Patients who wish to change treatment before the study ends will be withdrawn from the study.

During the study the investigators will ask patients to complete some standard questionnaires that are normally used to score the degree of the incontinence and to assess bowel symptoms.: These will be completed at the hospital during the standard clinic consultation, both before patients start the treatment and after having completed the treatment course.

ELIGIBILITY:
Inclusion Criteria:

* Passive or mixed faecal incontinence.
* Minimum two or more episodes of faecal incontinence per week as assessed by prospectively collected bowel diaries.
* Failed biofeedback, pelvic floor physiotherapy or other medical management.
* Able to self- administer the Renew™ Anal Insert.
* Competent and willing to fill in questionnaires and attend clinics throughout the study.
* Patient must be able to comprehend and informed consent prior to enrolment in the study.

Exclusion Criteria:

* Pregnancy.
* Inability to given informed consent.
* Perianal sepsis.
* Rectal bleeding.
* Inflammatory bowel disease/ Proctitis.
* Rectal prolapse.
* Third or fourth-degree hemorrhoids.
* Anal stricture.
* Anal or Recto-vaginal fistula.
* Rectal surgery in the past 3 months.
* Known allergy to Silicone.
* Patients who are mentally or physically unable to comply with the protocol of the study.
* The presence of any other medical condition which, in the opinion of the Chief Investigator, deems the patient unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2018-08-11 (Actual); Study Completion 2018-09-11 (Actual)

PRIMARY OUTCOMES:
Renew vs PTNS treatment | 3 months
  A consecutive two weeks bowel diaries at 3 months follow up Use of PTNS or RENEW Frequency of episodes of faecal incontinence

SECONDARY OUTCOMES:
Pain | 3 months
  Five-point visual analog scale (VAS) from 0 to 10
Severity of incontinence | 3 months
  This will be measured using a single validated outcome measure valued in score (St Mark's faecal incontinence score): this measure in a grade from 0 to 4, the number of episodes of incontinence to solid stools, the number of episodes of incontinence to liquid stools, the number of episodes of incontinence to flatus (gas). It also measures in a grade from 0 to 4 the frequency of the use of pads and the frequency of use constipating medicines. The sum of the numbers will give a final score which will be used as method to measure the severity of incontinence.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jorge JM, Wexner SD. Etiology and management of fecal incontinence. Dis Colon Rectum. 1993 Jan;36(1):77-97. doi: 10.1007/BF02050307. PMID 8416784
- [Background] Norton C, Kamm MA. Anal plug for faecal incontinence. Colorectal Dis. 2001 Sep;3(5):323-7. doi: 10.1046/j.1463-1318.2001.00257.x. PMID 12790954
- [Background] Horrocks EJ, Chadi SA, Stevens NJ, Wexner SD, Knowles CH. Factors Associated With Efficacy of Percutaneous Tibial Nerve Stimulation for Fecal Incontinence, Based on Post-Hoc Analysis of Data From a Randomized Trial. Clin Gastroenterol Hepatol. 2017 Dec;15(12):1915-1921.e2. doi: 10.1016/j.cgh.2017.06.032. Epub 2017 Jun 21. PMID 28647458
- [Background] Segal JP, Leo CA, Hodgkinson JD, Cavazzoni E, Bradshaw E, Lung PFC, Ilangovan R, Vaizey CJ, Faiz OD, Hart AL, Clark SK. Acceptability, effectiveness and safety of a Renew(R) anal insert in patients who have undergone restorative proctocolectomy with ileal pouch-anal anastomosis. Colorectal Dis. 2019 Jan;21(1):73-78. doi: 10.1111/codi.14422. Epub 2018 Oct 8. PMID 30218632
- [Derived] Leo CA, Thomas GP, Hodgkinson JD, Leeuwenburgh M, Bradshaw E, Warusavitarne J, Murphy J, Vaizey CJ. Randomized Pilot Study: Anal Inserts Versus Percutaneous Tibial Nerve Stimulation in Patients With Fecal Incontinence. Dis Colon Rectum. 2021 Apr 1;64(4):466-474. doi: 10.1097/DCR.0000000000001913. PMID 33399411